CLINICAL TRIAL: NCT00694538
Title: Efficacy of Interferential Laser Therapy in Pain Reduction in Shoulder Musculoskeletal Pathologies.
Brief Title: Efficacy of Interferential Laser Therapy in Shoulder Pain
Acronym: PI070046
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: MONTES-MOLINA, RAMON, HOSPITAL RAMON Y CAJAL- IMSALUD.
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PI070046; PI 070046
Record Dates: First submitted 2008-05-29; First posted 2008-06-10 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Shoulder Musculoskeletal Disorders
Keywords: Interferential laser therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 100 patients are being treated with a single laser beam over pain area.
  Interventions: Device: Interferential Laser therapy
- 2 (Experimental): 100 patients are being treated with interferential laser from two independent sources
  Interventions: Device: Interferential Laser therapy

INTERVENTIONS:
Device: Interferential Laser therapy — Two GaAlAs laser (810 nm, 100mW)were used. In the interferential laser treatment, two probes were simultaneously applied. In the conventional laser group, only one probe was switched on. Laser was applied at five points over the pain area. The laser emission mode was continuous with an energy dose of 6 joules per point and session, a power density of 1.09 w/cm2 and an irradiation time per point of 60 s. The average output power was 100 mW and the total energy dose delivered in a patient session was 30 J. Every treatment was along 15 sessions. Hence, the accumulated energy delivered on the whole was 450 Joules for the conventional group of patients (using one beam) and 900 Joules for the interferential one (using two beams).
  Other Names: Interference Laser Therapy.; Device Brand Name: Laser Sys. Stim 540(Mettler Electronics).; SN: 105XLS147 (first laser) and 105XLS148 (second laser).

SUMMARY:
The purpose of this study is to determine the advantages of the interferential laser therapy in shoulder pain reduction compared with the conventional low level laser therapy modality.

DETAILED DESCRIPTION:
The spatiotemporal superposition of two independent and opposite beams of laser generates a constructive interference pattern that increases the therapeutic effects in the irradiated tissue. Patients diagnosed of shoulder pain from different musculoskeletal disorders will received conventional or interferential laser therapy. This is a comparative, randomized and double - blind clinical study. Two identical equipments of near infrared laser therapy will be used. Number of sessions: 15. Frequency of the sessions: daily. Irradiation technique: manual, contact and punctual.Pain will be evaluated by visual analog scale (VAS) at rest and during analytical shoulder movements (abduction, adduction, internal rotation, external rotation, flexion, extension) and by means of a pain and disability index (SPADI). Evaluations will take place at pre and post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Acute or chronic pain from musculoskeletal origin
* Age between 18 and 70 years

Exclusion Criteria:

* Brachial plexus palsy
* Neurological diseases
* Pacemakers
* Shoulder pain from cervical pathology
* Osteosynthesis material
* Fibromyalgia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Pain will be evaluated by visual analog scale (VAS) at rest and during analytical shoulder movements. | Five minutes

SECONDARY OUTCOMES:
Shoulder Pain Disability Index (SPADI) | ten minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Montes-Molina, PT, Principal Investigator — Hospital Ramon y Cajal
Locations (1):
- Hospital Ramon y Cajal, Madrid, Madrid, Spain

REFERENCES:
- [Background] Montes-Molina R, Madronero-Agreda MA, Romojaro-Rodriguez AB, Gallego-Mendez V, Prados-Cabiedas C, Marques-Lucas C, Perez-Ferreiro M, Martinez-Ruiz F. Efficacy of interferential low-level laser therapy using two independent sources in the treatment of knee pain. Photomed Laser Surg. 2009 Jun;27(3):467-71. doi: 10.1089/pho.2008.2315. PMID 19405858
- [Derived] Montes-Molina R, Prieto-Baquero A, Martinez-Rodriguez ME, Romojaro-Rodriguez AB, Gallego-Mendez V, Martinez-Ruiz F. Interferential laser therapy in the treatment of shoulder pain and disability from musculoskeletal pathologies: a randomised comparative study. Physiotherapy. 2012 Jun;98(2):143-50. doi: 10.1016/j.physio.2011.02.007. Epub 2011 May 28. PMID 22507365